CLINICAL TRIAL: NCT06868927
Title: Targeted Decision Making In Renal Cell Carcinoma Relying on a Radiogenomics Translational Platform
Acronym: TARGET-RCC
Status: Not yet recruiting | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Umberto Capitanio, Group Leader Renal Cancer Lab, IRCCS San Raffaele
Other Study IDs: TARGET-RCC
Record Dates: First submitted 2025-02-26; First posted 2025-03-11 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-01

CONDITIONS: Renal Tumors
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This project aims to provide an accurate strategy to guide the decision making relying on tumor biopsies using standard histology, immunohistochemistry (IHC), spatial transcriptomics, genomics combined with Magnetic Resonance Imaging (MRI) and radiomics. Moreover, the investigators will explore potential markers indicative of response to systemic agents or ablative therapy.

ELIGIBILITY:
Inclusion Criteria:

* Presence of a renal mass up to 4 cm
* Adult > 18 years
* Candidate to renal surgery
* Informed consent signed

Exclusion Criteria:

* Contraindication for MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: subjects with a renal tumor up to 4 cm and candidates for surgery
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-05-15 (Estimated); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
accuracy of multiparametric preoperative MRI | At final pathological assessment , at least 1 month after surgery
  Detection of "Unfavourable outcome" is defined as the presence of at least one of the following pathological characteristics:
  * High grade tumor (G3 or G4)
  * Not-organ confined disease (pT3 and or pT4 and/or LNI)
  * Sarcomatoid features